CLINICAL TRIAL: NCT06345326
Title: Comparison of the Clinical Effectiveness of Repeated Ultrasound-guided Greater Occipital Nerve Blocks and Greater Occipital Nerve Pulse RF in the Treatment of Migraine
Brief Title: Greater Occipital Nerve Block Versus Pulse Radiofrequency in Migraine
Acronym: GON-B/PRF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Collaborators: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Dr. Ülkü Sabuncu, M.D., Ankara City Hospital Bilkent
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E1-22-3155
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Migraine
Keywords: migraine; greater occipital nerve block; pulse radiofrequency
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Prospective observational
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repeated greater occipital nerve block (Experimental): In this arm, all the participiants will receive ultrasound guided greater occipital nerve block for a week, for 4 weeks with ultrasound guidiance at the level C2
  Interventions: Other: Greater occipital nerve block
- Greater occipital nerve pulse radiofrequency (Experimental): In this arm, all the participiants will receive ultrasound guided greater occipital nerve pulse radiofrequency with ultrasound guidiance at the level C2
  Interventions: Other: Greater occipital nerve block

INTERVENTIONS:
Other: Greater occipital nerve block — The nerve block will be done by ultrasound guidiance at the C2 level with a 22 gauge 5 cm needle inplane direction. The pulse radiofrequency will be done as defined with a radiofrequency cannula- 5 cm with an active tip of 2mm.
  Other Names: Pulse radiofrequency

SUMMARY:
The aim of the study is to evaluate the clinical efficacy of the repeated greater occipital nerve(GON) blokcs with GON pulse radiofreaquency (PRF)

DETAILED DESCRIPTION:
The nerve blocks will be performed at the Cervical-2 (C2) level with ultrasound guidance.Also , the PRF will be done as above proximally.

ELIGIBILITY:
Inclusion Criteria:

* ICHD- migraine with minimum 4 attacks
* no benefit with proflactic therapies

Exclusion Criteria:

* primary headhache other than migraine according to ICHD
* the change of medical teatment of migrane in last 1 month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
NRS | Before the application then every month following the intervention for 3 months
  Numeric rating scala

SECONDARY OUTCOMES:
Complications | Before the application then every month following the intervention for 3 months
  vertigo, dizzines, hypotension , bleeding, local pain ect.
the frequency of headhache | Before the application then every month following the intervention for 3 months
  how many times the headhache occured

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital Bilkent, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided